CLINICAL TRIAL: NCT05529446
Title: Effect of Combination Therapy on Knee Osteoarthritis Pain in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Madonna Noshi Welson Aiad, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003571
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Non Specific Knee Osteoarthritis Pain
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): This group will consist of twenty women with mild to moderate osteoarthritis suffering from pain. These women will perform strengthening exercises in addition to combination therapy 10 minutes for each session, 3 times per week, for 3 weeks.
  Interventions: Device: Combination therapy (CT)
- control (Sham Comparator): This group will consist of twenty women with mild to moderate osteoarthritis suffering from pain.These women will perform the same strengthening exercises as intervention group and receive sham combination therapy 10 minutes for each session, 3 times per week, for 2 weeks.
  Interventions: Device: Combination therapy (CT)

INTERVENTIONS:
Device: Combination therapy (CT) — Two therapeutic modalities at the same site is described as combination therapy (CT). The most commonly used CT is US & TENS where this approach was effective in pain modulation

SUMMARY:
the aim of this study is to investigate the efficacy of Combination Therapy on Knee Osteoarthritis Pain in Postmenopausal Women

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common musculoskeletal condition affecting the quality of life of older adults. The prevalence of OA is very high 45% in females in comparison to males, especially after menopause due to the hormonal changes. In the physical therapy practice, therapeutic ultrasound (US) is one of the most frequently applied electrotherapeutic modalities in orthopedics physiotherapy. Simultaneous application of two therapeutic modalities at the same site is described as combination therapy (CT). The most commonly used CT is US & Transcutaneous neuromuscular electrical stimulation (TENS )where this approach was effective in pain modulation .The use of combination therapy is highly preferable because of the advantageous effect both electro-therapy and ultrasound provide simultaneously. There are no current studies on using combination therapy in the treatment of pain in mild to moderate knee osteoarthritis in post-menopausal women and we don't know the proper treatment dose.The study is designed as a prospective, randomized, pre-posttest, controlled trial.where we have two groups Intervention group and control. the intervention group will recieve strengthening exercises in addition to combination therapy 10 minutes for each session, 3 times per week, for 3 weeks.The Control group will recieve the same strengthening exercises as intervention group and sham combination therapy 10 minutes for each session, 3 times per week, for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Forty women who suffer pain out of mild to moderate knee osteoarthritis
* Their age will range from 55 to 65
* At least one year after last menstruation.
* Their BMI will be ranged from 25 to 35 kg/m2

Exclusion Criteria:

* Neurological disorders.
* Cardiovascular disorders.
* Severe knee osteoarthritis
* Areas of the body where cancerous lesions exist.
* Any skin impairment at site of application as inflammation, lesion, wounds, infection and swelling.
* Pacemaker and any metallic implants.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Knee Range Of Motion | up to four weeks
  electronic goniometer it measures range of motion objectively assess ROM for extremities and digits

SECONDARY OUTCOMES:
activity of daily living | up to four weeks
  Western Ontario and McMaster universities arthritis index (WOMAC) It will be used to measure activities of daily living, functional mobility gait, general health and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Madonna Noshi Welson Aiad, Cairo, Egypt